CLINICAL TRIAL: NCT06074848
Title: Transcranial Direct Current Stimulation as a Strategy for the Management of Disorders Generated by COVID-19: a Multicentric Study.
Brief Title: tDCS in the Management of Post-COVID Disorders
Acronym: tDCS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: São Paulo State University (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Investigador principal, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS_COVID
Record Dates: First submitted 2023-08-26; First posted 2023-10-10 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Long COVID
Keywords: Long COVID; Post-Acute COVID-19 Syndrome; Fatigue; Pain; Cognitive Dysfunction; Depression; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; Pain; Cognitive Dysfunction; Depression | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pain/fatigue tDCS real (Experimental): tDCS will be applied for 30 minutes (2 mA; 0.057 mA/cm²) during motor training. The anode will be positioned in the area referring to the left motor cortex (C3). The cathode will be positioned in the contralateral supraorbital region.
  Motor Training: the participant will be positioned on the mat where the initial 5 minutes will be warmed up with the target heart rate maintained at 50-60% of the maximum heart rate. The treadmill speed must be adjusted to keep the HR within the pre-established target range. At 5 minutes, Borg scale values, treadmill speed and HR should be recorded. The central 20 minutes will be considered the main part. For this, the target HR must be maintained between 64-76% of the maximum HR. Every 5 minutes (minutes 10, 15, 20 and 25) the values of the Borg scale, treadmill speed and HR must be recorded. In the final 5 minutes, the target HR must be kept below 60% of the maximum HR. Totaling 30 minutes of training on the treadmill.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Motor Training
- Pain/fatigue tDCS sham (Sham Comparator): tDCS will be applied for 30 seconds (2 mA; 0.057 mA/cm²) during motor training. The anode will be positioned in the area referring to the left motor cortex (C3). The cathode will be positioned in the contralateral supraorbital region.
  Motor Training: the participant will be positioned on the mat where the initial 5 minutes will be warmed up with the target heart rate maintained at 50-60% of the maximum heart rate. The treadmill speed must be adjusted to keep the HR within the pre-established target range. At 5 minutes, Borg scale values, treadmill speed and HR should be recorded. The central 20 minutes will be considered the main part. For this, the target HR must be maintained between 64-76% of the maximum HR. Every 5 minutes (minutes 10, 15, 20 and 25) the values of the Borg scale, treadmill speed and HR must be recorded. In the final 5 minutes, the target HR must be kept below 60% of the maximum HR. Totaling 30 minutes of training on the treadmill.
  Interventions: Behavioral: Motor Training
- Cognitive deficit and depressed mood tDCS real (Experimental): tDCS will be applied for 30 minutes (2 mA; 0.057 mA/cm²) during cognitive training. For volunteers with symptoms of depressed mood and/or cognitive impairment, the anode will be positioned in the area of the left dorsolateral prefrontal cortex (F3) and cognitive training will be performed. The cathode will be positioned in the contralateral supraorbital region.
  Cognitive Training: For cognitive training, performed during tDCS, a n-Back task will be performed online in the PsyToolkit (https://www.psytoolkit.org/). A previous study demonstrated the benefit of tDCS when combined with this cognitive training on working memory learning curves.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive Training
- Cognitive deficit and depressed mood tDCS sham (Sham Comparator): tDCS will be applied for 30 seconds (2 mA; 0.057 mA/cm²) during cognitive training. For volunteers with symptoms of depressed mood and/or cognitive impairment, the anode will be positioned in the area of the left dorsolateral prefrontal cortex (F3) and cognitive training will be performed. The cathode will be positioned in the contralateral supraorbital region.
  Cognitive Training: For cognitive training, performed during tDCS, a n-Back task will be performed online in the PsyToolkit (https://www.psytoolkit.org/). A previous study demonstrated the benefit of tDCS when combined with this cognitive training on working memory learning curves.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS deliver low-intensity electrical currents (2 mA) through electrodes placed on the scalp. It is used to influence brain function, modulating the neuronal activity in specific areas, in a non-invasive way, as the stimulation may not be perceived sensorially due to the low intensity. In some cases, it can provide mild tingling and bring minimal discomfort. It has the ability to increase or decrease the cortical excitability of neurons, influencing the polarization of neuronal membranes, with the anodal pole (positive) facilitating depolarization that results in increased neuronal excitability in the area, and the cathodal pole (negative) promoting a hyperpolarization of the neuronal resting membrane potential that reduces cortical excitability, used to inhibit activity in a particular cortical area.
  Other Names: non-invasive brain stimulation, neuroConn (Germany)
  Arms: Cognitive deficit and depressed mood tDCS real; Pain/fatigue tDCS real
Behavioral: Motor Training — Motor training will be performed on the treadmill with the speed respecting the limits of the patient's maximum heart rate. To determine the maximum heart rate, the calculation must be performed: maximum heart rate = 208 - (0.7*age). For participants who use beta-blockers, the following formula will be used: maximum heart rate = 164 - (0.7*age). Just for the arms of fatigue and pain.
  Arms: Pain/fatigue tDCS real; Pain/fatigue tDCS sham
Behavioral: Cognitive Training — an n-Back task will be performed online at PsyToolkit (https://www.psytoolkit.org/). Just for the arms of cognitive impairment and depressed mood.
  Arms: Cognitive deficit and depressed mood tDCS real; Cognitive deficit and depressed mood tDCS sham

SUMMARY:
Different physical and mental morbidities such as pain, fatigue, depressed mood and cognitive impairment can be triggered by coronavirus infection. Transcranial direct current stimulation (tDCS), an easy-to-apply, non-pharmacological and safe technique, has been used to attenuate these symptoms caused by other diseases, and, therefore, it is expected that it can also attenuate them when generated by COVID-19. It is known that the persistent inflammatory state observed after COVID-19 would be related to the progression of these negative symptoms. As non-invasive brain stimulation can also attenuate acute and persistent inflammation, it can be estimated that tDCS can be a useful tool to recover immune function and reduce post-COVID-19 morbidity.

DETAILED DESCRIPTION:
The aim of this study is to investigate if Direct Current Electrical Stimulation (tDCS) associated with motor and/or cognitive training is capable of reducing neuropsychiatric symptoms, as well as immune changes induced in COVID-19.

Volunteers will be randomized and allocated into four groups (Fatigue; Pain; Cognitive deficit and Depressed mood) and each group will be divided into two subgroups: 1) real tDCS + motor or cognitive training; and, 2) sham tDCS + motor or cognitive training according to each outcome. The volunteers will be evaluated in two aspect: immunometabolic evaluation (i) and clinical assessment (ii). The measures will pe performed in three moments: baseline (session 1); 72 hours after the last intervention (session 12) and follow up - 15 days after the last intervention (session 13).

(i) The immunometabolic evaluation will start with the participant's blood collection, after fasting for 8-12 hours, without having practiced intense physical activity and without drinking alcohol in the 24 hours prior to the collect. The blood will be allocated in 10 vacutainer tubes of 5ml containing EDTA for plasma separation, in 2 dry vacutainer tubes of 5ml for serum separation and 1 vacutainer tube of 5ml containing fluoride. In particular, 1 dry tube must rest for 1h, for subsequent BDNF analysis. 2 serum tubes, 2 plasma tubes and 1 fluoride tube should be centrifuged at 3,500 rpm for 15 minutes at 4°C, and the samples should be stored at -80°C for later analysis and the other fresh plasma tubes used (up to 2 hours after collection) for whole blood and PBMC stimuli.

Stimulation of whole blood with LPS, culture of peripheral blood mononuclear cells (PBMC), assessment of oxidative stress, assessment of adenine and LPS purine levels in plasma, analysis of immunophenotyping and apoptosis by flow cytometry, assessment of expression of purinoreceptors, mitochondrial assays in monocytes and T lymphocytes, evaluation of the generation of reactive oxygen species and quantification of several mediators by ELISA.

(ii) The clinical assessment will be performed using the following outcome measures:

COVID clinical situation - IInitially, modules 1 and 2 of the Case Report Form - CRF (Pcovid frameost COVID-19 CRF) of the Pan American Health Organization (PAHO) will be completed. Where module 1 comprises demographic data and clinical information related to the acute episode of COVID-19 and module 2 includes questions related to vaccination, occupational and functional status of the volunteer.

Fatigue - The Modified Impact of Fatigue Scale (MFIS) contains 21 items that analyze cognitive, physical and psychosocial issues in relation to fatigue, assessing the impact that is caused in the patient's life.

Pain - Brief Pain Inventory (BPI) assesses pain severity, impact of pain on daily function, pain location, pain medications, and amount of pain relief in the last 24 hours and last week; Visual Analog Scale (VAS) consists of a ruler numbered from 0 to 10 and divided into three parts, light, moderate and severe, with visual aid to facilitate the measurement of the patient's pain intensity.

Cognitive deficit - Montreal Cognitive Assessment (MoCA) instrument that quickly identifies cognitive declines in patients; FAS Test is a Verbal Fluency Test - Phonological Fluency Test that assesses verbal learning and the ability to produce words verbally; Random Number Generator (RNG test) assesses language and executive function; Digit span that will be used to assess the ability to focus, maintain attention, and mental manipulation. In the follow up, the CFL-test will be added to a verbal fluency test.

Depressed mood - Hospital Anxiety and Depression Scale (HADS) measures symptoms of anxiety and depression and consists of 14 items, seven for the anxiety subscale (HADS-Anxiety) and seven for the depression subscale (HADS-Depression); Brunel Mood Scale (BRUMS) used to quickly measure the patient's mood state.

Level of physical activity - The short version of IPAQ will be performed to identify if the volunteer has a life with active physical activities. It makes it possible to estimate the weekly time used for physical activities.

Vital signs - at the end of the scales, the signs of each patient will be measured: blood pressure, heart rate, respiratory rate and peripheral O2 saturation, parameters used to verify the hemodynamic status of the volunteer.

State of strength and effort - the handgrip strength test and perception of effort performed with the dynamometer will be used, quantitatively indicating the muscle strength of the hand and forearm.

Exercise capacity - the functional capacity and aerobic resistance of the participant will be evaluated through the 6-minute walk test. The test measures the distance that the volunteer covers in a period of 6 minutes walking at a stable speed.

At the end, a questionnaire of adverse effects of the evaluation will be carried out, containing information regarding any discomfort felt during the evaluation.

The intervention process will be carried out with Transcranial Direct Current Stimulation which will be applied for 30 minutes (2 mA; 0.057 mA/cm²) during motor or cognitive training. For symptoms of pain and/or fatigue, the anode will be positioned in the area referring to the left primary motor cortex (C3, according to the EEG positioning system). For symptoms of depressed mood and/or cognitive impairment, the anode will be positioned in the area of the left dorsolateral prefrontal cortex (F3). In both situations, the cathode will be positioned in the contralateral supraorbital region. In sham tDCS, the same parameters and setup as the real stimulation will be used, however, the application time will be 30 seconds, but the electrodes will be maintained for 30 minutes.

In motor training, the treadmill training protocol will last a total of 30 minutes and will be carried out during the application of tDCS. After positioning the tDCS electrodes, a cardiac monitor will be positioned on the individual to control HR. Before starting the protocol on the treadmill, the values of the perceived exertion scale (Borg) and HR should be noted.

Initially, the target HR for each part of the intervention will be determined. The formula by Tanaka et al., (2001) will be used to determine the maximum HR, with maximum HR = 208 - (0.7*age). For participants who use beta-blockers, the formula by Brawner et al., (2004) will be used, with maximum HR = 164 - (0.7*age).

The initial five minutes will be a warm-up. To achieve this, the target HR must be maintained at 50-60% of the maximum HR. The speed of the treadmill must be adjusted to maintain the HR within the pre-established target range. At five minutes, the Borg scale values, treadmill speed and HR must be noted. The central 20 minutes will be considered as the main part. To achieve this, the target HR must be maintained at 64-76% of the maximum HR. If the participant chooses to stop the treadmill session, the treadmill must be turned off and the participant must remain seated until the end of the tDCS application.

For cognitive training, carried out during tDCS, an n-Back task will be performed online in PsyToolkit (https://www.psytoolkit.org/). For a benefit on working memory learning curves. Performed for the outcomes of cognitive impairment and depressed mood. During the test, the volunteer will have to indicate which letter was projected by the application two letters ago. The system will show one letter followed by another, the volunteer must press the "space" key on the computer keyboard when the letter that was shown in the two positions above reappears.

The study will be carried out simultaneously in two research centers in Brazil: Laboratory of Applied Neuroscience (LANA), Federal University of Pernambuco (UFPE), Pernambuco, Brazil and at the Department of Physical Education, Faculty of Science and Technology - Campus Presidente Prudente (FCT/UNESP), São Paulo, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID-19 (>3 months)
* The presence of at least one of the following symptoms, after diagnosed SARS-COV-2 infection:

Persistent pain Fatigue Depressed mood Cognitive impairment

Exclusion Criteria:

* Hemodynamic instability
* Historic of use or abuse of drugs or alcohol
* Use of medications that may interfere with the study results (anti-inflammatories and antibiotics)
* Metallic implant in skull and face
* Implant in the central nervous system
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-28 (Estimated)

PRIMARY OUTCOMES:
Fatigue - Modified Fatigue Impact Scale (MFIS) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  The MFIS is a scale that contains 21 items that analyze cognitive, physical and psychosocial issues. The physical domain allows scores from 0 to 36, the cognitive domain from 0 to 40 and the psychosocial domain from 0 to 8. The total MFIS score is given by the sum of the three domains and varies from 0 to 84 points. Values below 38 correspond to the absence of fatigue, and above this value, the higher the score, the greater the individual's degree of fatigue.
Pain measure - Brief Pain Inventory (BPI) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  assesses severity of pain, impact of pain on daily functions, location of pain, analgesics, and amount of pain relief in the past 24 hours and past week on an 11-point scale ranging from 0 (no pain/no interference) to 10 (the worst possible). Including a body diagram to assess the location of pain (item 2), scores range from 0 to 10 and are calculated as the average of the total items. A high score represents a high pain intensity or pain interference
Pain measure - Visual Analog Scale (VAS) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  consiste em uma régua numerada de 0 a 10 e dividida em três partes, leve, moderada e intensa, com auxílio visual para facilitar a mensuração da intensidade da dor do paciente.
Cognitive deficit - Montreal Cognitive Assessment Instrument (MoCA) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  quickly identifies cognitive declines in patients with a maximum score of 30 (points), evaluates eight cognitive domains: 1. Executive function: with the Trail Making Test B (adapted - 1 point), phonemic verbal fluency (1 point) and abstraction verbal (2 points). 2. Visual-spatial ability: drawing the clock (3 points) and copying the cube (1 point). 3. memory: delayed recall of words 5 minutes (5 points). 4. Attention/5. Concentration/6. Working memory: digit memory (forward sense - 1 point), digit memory (backward sense - 1 point), sustained attention task (target detection - 1 point) and serial subtraction of 7 (3 points). 7. Language: naming 3 unfamiliar animals (3 points), repetition of 2 syntactically complex sentences - phonemic verbal fluency (above - 2 points). 8. Orientation: temporal (4 points) and spatial (2 points). It has a total score of 30 points. The cutoff score is 26 points, indicating the presence of cognitive deficit. Score above said is considered normal.
Cognitive deficit - FAS Test | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  is a Verbal Fluency Test/Phonological Fluency Test that assesses verbal learning and the ability to produce words verbally. The total score is given by adding up all correct words starting with the three letters.
Cognitive deficit - CFL Test | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  is a Verbal Fluency Test/Phonological Fluency Test that assesses verbal learning and the ability to produce words verbally. The total score is given by adding up all correct words starting with the three letters.
Cognitive deficit - Random Number Generator | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  Assesses language and executive function. Numbers are produced randomly when a previously recorded sound signal is heard. You must speak numbers from 1 to 10 without speaking sequences.
Cognitive deficit - Digit span | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  Used to assess the ability to focus, maintain attention, mental manipulation and memory. It consists of repeating the numbers said by the evaluator, where in the first phase they will be said in direct order (16 points) and in the second phase in reverse order (14 points). Together they add up to a maximum score of 30 points.
Depressed mood - Hospital Anxiety and Depression Scale (HADS) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  measures symptoms of anxiety and depression divided into an anxiety subscale (HADS-Anxiety) and a depression subscale (HADS-Depression). Each question has a variable score from zero to four points, with 14 questions in total. From 0 - 7 points indicates anxiety and depression unlikely; 8 - 11 points indicate possible anxiety and depression and 12 - 21 points indicate probable anxiety and depression.
Depressed mood - Brunel Mood Scale (BRUMS) | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  Used to quickly measure a patient's mood using six subscales: tension, depression, anger, vigor, fatigue and confusion. It contains 24 questions that must be evaluated according to a scale of 0 to 4 points, each subscale has a score that can vary from 0 - 16.

SECONDARY OUTCOMES:
COVID clinical situation | pre-intervention
  It will be carried out using the Case Report Form - CRF (Post COVID-19) from the Pan American Health Organization (PAHO). Using the first two modules, module 1 comprises demographic data and clinical information related to the acute episode of COVID-19 and module 2 includes questions related to vaccination, occupational and functional status of the volunteer. Based on these questionnaires, it is possible to identify the patient's status in their episodes of contagion with COVID-19 and the degree of support that was needed in each case, as well as the main symptoms and characteristics of the case.
Level of physical activity | pre-intervention
  The short version of IPAQ will be performed to identify if the volunteer has a life with active physical activities. It makes it possible to estimate the weekly time used for physical activities.
State of strength and effort | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  the handgrip strength test and perceived exertion performed with the dynamometer will be used to quantitatively indicate the muscle strength of the hand and forearm and to assess the level of effort exerted through the BORG scale.
Exercise capacity - 6-minute walk test | pre-intervention, 72 hours after the last intervention and 15 days after completion.
  the participant's functional capacity and aerobic resistance will be evaluated through the 6-minute walk test. The test measures the distance that the volunteer covers in a period of 6 minutes walking at a steady speed.
Immunometabolic evaluation | pre-intervention and 72 hours after the last intervention
  will begin with the participant's blood collection. Stimulation of whole blood with LPS, culture of peripheral blood mononuclear cells (PBMC), evaluation of oxidative stress, evaluation of adenine and purine LPS levels in plasma, analysis of immunophenotyping and apoptosis by flow cytometry, evaluation of expression of purinoreceptors, mitochondrial assays in monocytes and T lymphocytes, evaluation of the generation of reactive oxygen species and quantification of several mediators by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Lopes, graduation, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Lívia Shirahige, PhD, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Bárbara Sousa, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Ana Cecília, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Adriana Baltar, PhD, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Rodrigo De Mattos, Master, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Gabriel Barreto, Master, Study Chair — Laboratory of Applied Neuroscience, Federal University of Pernambuco; Fábio Santos de Lira, PhD, Study Chair — Department of Physical Education, Faculty of Science and Technology - Presidente Prudente Campus; Fabrício Oliveira Souto, PhD, Study Chair — Universidade Federal de Pernambuco; Kátia Monte-Silva, PhD, Study Director — Laboratory of Applied Neuroscience, Federal University of Pernambuco
Locations (2):
- Brazil (2):
  - Applied Neuroscience Laboratory-LANA, Recife, Pernambuco
  - Department of Physical Education, Faculty of Science and Technology, Presidente Prudente, São Paulo

REFERENCES:
- See also: Choi, Hyo Jung, Dong Young Lee, et al. 2014. "A Normative Study of the Digit Span in an Educationally Diverse Elderly Population." Psychiatry Investigation 11 (1): 39-43. — https://pubmed.ncbi.nlm.nih.gov/24605122/
- See also: Dorneles, Gilson P., Paula C. Teixeira, et al. 2022. "Alterations in CD39/CD73 Axis of T Cells Associated with COVID-19 Severity." Journal of Cellula — https://pubmed.ncbi.nlm.nih.gov/35754396/
- See also: Lira, Pereira, and Guerra Minuzzi. "Functions in Adult Patients with Mild to Moderate SARS-CoV-2 Infections-A Protocol for an Observational Prospective Follow-Up Investigation: Fit-COVID-19." International Journal of High Risk Behaviors & Addict. 2021 — https://observatorio.fm.usp.br/handle/OPI/48228
- See also: Postiga, Isabelle A. L., Paula C., et al. "Systemic Redox Imbalance in Severe COVID-19 Patients." Cell Biochemistry and Function, August. 2022. — https://pubmed.ncbi.nlm.nih.gov/35980161/
- See also: Romão PR, Teixeira PC, Schipper L, et al. Viral load is associated with mitochondrial dysfunction and altered monocyte phenotype in acute severe SARS-CoV-2 infection. Int Immunopharmacol. 2022 Jul;108:108697. doi: 10.1016/j.intimp.2022.108697. — https://pesquisa.bvsalud.org/global-literature-on-novel-coronavirus-2019-ncov/resource/pt/covidwho-1739816
- See also: Rossini, PM et al. 2015. "Non-Invasive Electrical and Magnetic Stimulation of the Brain, Spinal Cord, Roots and Peripheral Nerves: Basic Principles and Procedures for Routine Clinical and Research Application. An Updated Report from an IFCN Committee — https://pubmed.ncbi.nlm.nih.gov/25797650/
- See also: Scarpina, Federica, and Sofia Tagini. 2017. "The Stroop Color and Word Test." Frontiers in Psychology 8 (April): 557. — https://pubmed.ncbi.nlm.nih.gov/28446889/
- See also: Teixeira PC, Dorneles GP, Santana Filho PC, et al. Increased LPS levels coexist with systemic inflammation and result in monocyte activation in severe COVID-19 patients. Int Immunopharmacol. 2021 Nov;100:108125. doi: 10.1016/j.intimp.2021.108125. — https://pubmed.ncbi.nlm.nih.gov/34543980/
- See also: Versace, Viviana, Luca Sebastianelli, et al. 2021. "Intracortical GABAergic Dysfunction in Patients with Fatigue and Dysexecutive Syndrome after COVID-19." Clinical Neurophysiology: Official Journal of the Int Federation of Clinical Neurophysiol — https://pubmed.ncbi.nlm.nih.gov/33774378/
- See also: Yang, L., Liu, S., Liu, J. et al. COVID-19: immunopathogenesis and Immunotherapeutics. Sig Transduct Target Ther 5, 128 (2020) — https://doi.org/10.1038/s41392-020-00243-2
- See also: Organização Pan-Americana da Saúde. Plataforma Clínica Global da COVID-19 Ficha Clínica (Case Report Form - CRF) para quadro pós-COVID (Post COVID-19 CRF). OPAS-W/BRA/PHE/COVID-19/21-0025 (2021). — https://cdn.who.int/media/docs/default-source/3rd-edl-submissions/who_crf_postcovid_feb9_2021.pdf